CLINICAL TRIAL: NCT05745311
Title: A Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Phase II Clinical Trial Evaluating the Efficacy and Safety of the KPCXM18 Injection in Patients With Acute Ischemic Stroke.
Brief Title: Study of the KPCXM18 Injection for Treatment of Acute Ischemic Stroke
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kunming Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KPCXM18/C201
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low-dose group （The KPCXM18 injection） (Experimental): Intravenous infusion of 20 mg twice daily at intervals of 12±2 hours for 10 days.
  Interventions: Drug: The KPCXM18 injection
- middle-dose group （The KPCXM18 injection） (Experimental): Intravenous infusion of 60 mg twice daily at intervals of 12±2 hours for 10 days.
  Interventions: Drug: The KPCXM18 injection
- high-dose group （The KPCXM18 injection） (Experimental): Intravenous infusion of 100 mg twice daily at intervals of 12±2 hours for 10 days.
  Interventions: Drug: The KPCXM18 injection
- Placebo (Placebo Comparator): Intravenous infusion twice a day with an interval of 12±2 hours for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: The KPCXM18 injection — Intravenous infusion
  Arms: high-dose group （The KPCXM18 injection）; low-dose group （The KPCXM18 injection）; middle-dose group （The KPCXM18 injection）
Drug: Placebo — Intravenous infusion
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, parallel, placebo-controlled trial design to evaluate the efficacy and safety of the KPCXM18 injection at different doses for the treatment of acute ischemic stroke and its PK/PD characteristics in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years old (including 18 years old and 80 years old), male or female;
2. Diagnosed with acute ischemic stroke according to the "Chinese guidelines for the diagnosis and treatment of acute ischemic stroke 2018";
3. The time from the last normal behavior to the time of initiation of the drug infusion ≤ 48 hours. For stroke after waking up or when the time of symptom onset cannot be accurately obtained due to aphasia, consciousness disorder, and other reasons, the time of onset should take the last time the patient showed normally as standard;
4. The patients who first attacked, or the patients who had a good prognosis after the last attacked ( mRS score was ≤1 before the onset of the disease );
5. During the screening period, 4 points ≤ NIHSS score ≤ 24 points, and the sum of NIHSS fifth upper limb and sixth lower limb score ≥2 points;
6. The subject or his guardian is aware of the study, and if the subject or his guardian is unable to read, the impartial witness reads the informed consent form and other written materials, witnesses the informed consent, voluntarily participates and signs the written informed consent.

Exclusion Criteria:

1. Patients with intracranial hemorrhagic diseases confirmed by head CT or MRI: hemorrhagic stroke, epidural hematoma, intracranial hematoma, ventricular hemorrhage, subarachnoid hemorrhage, etc;
2. Patients with disturbance of consciousness (NIHSS score Ia ≥2 points);
3. Patients who need or have undergone intravenous thrombolysis or endovascular interventional therapy (including endovascular mechanical thrombectomy, intravascular thrombus aspiration, arterial thrombolysis, angioplasty and stenting, etc.) or patients with arteriovenous bridging therapy after this onset;
4. Patients with malignant tumors, serious diseases of blood, digestion or other systems or diseases with bleeding tendencies (such as hemophilia, etc.), and the expected survival time is not more than 3 months;
5. Patients with a history of major surgery within 1 month before screening;
6. Patients with severe hypertension (systolic blood pressure ≥ 200 mmHg or diastolic blood pressure ≥110 mmHg) that cannot be controlled after treatment;
7. Patients with heart rate < 40 beats/min and/or ventricular rate > 120 beats/min; Patients with 2nd and 3rd degree heart blocks without pacemakers or other malignant arrhythmias; Patients with acute myocardial infarction, cardiac interventional therapy, or heart failure (grade III and IV according to NYHA) within the past 1 month;
8. Patients with severe liver function impairment, or ALT, AST > 2.0 times the upper limit of normal value (ULN);
9. Patients with severe renal impairment, or serum creatinine (Cr) > 1.5× ULN;
10. Patients who have used neuroprotective drugs (including commercially available edaravone, edaravone and dexborneol, nimodipine, gangliosides, piracetam, oxiracetam, butylphthalide, etc.) after the onset of this illness, as well as other traditional Chinese medicine labels containing the effect of treating acute ischemic stroke (cerebral infarction);
11. Patients with other psychiatric diseases and limb disorders, including severe mental disorders, dementia and other combined diseases that may affect neurological function tests;
12. Patients with a history of alcohol or drug abuse;
13. Patients with allergies, hypersensitivity to citicoline, KPCXM18 or excipients;
14. Pregnancy, lactation. or patients who have a family plan within 3 months of the first dose and who are unwilling to use contraception;
15. Patients who participated in or are currently participating in other clinical trials within 1 month prior to this study;
16. The investigator considers that patients are not suitable for clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in NIHSS score from baseline at day 10 after administration | day 10
  The National Institute of Health stroke scale(NIHSS) score ranging from 0-42. Higher score indicates worse function.

SECONDARY OUTCOMES:
Proportion of subjects with mRS score ≤ 1 at day 90±7 after administration | day 90±7
  The Modified Rankin Scale(mRS) score ranging from 0-5. Higher score indicates worse function.
Change in BI score from baseline at day 90±7 after administration | day 90±7
  The Barthel Index score ranges from 0 to 100, the higher scores mean a better outcome.
Change in EQ-5D score from baseline at day 90±7 after administration | day 90±7
Changes in NIHSS score from baseline on days 30±3 and 90±7 after administration | days 30±3 and 90±7
  The National Institute of Health stroke scale(NIHSS) score ranging from 0-42. Higher score indicates worse function.
Changes in mRS score from baseline on days 30±3 and 90±7 after administration | days 30±3 and 90±7
  The Modified Rankin Scale(mRS) score ranging from 0-5. Higher score indicates worse function.
The proportion of subjects whose NIHSS score improved by ≥4 points at days 10, 30±3 and 90±7 after administration | days 10, 30±3 and 90±7
  The National Institute of Health stroke scale(NIHSS) score ranging from 0-42. Higher score indicates worse function.
Proportion of subjects with recurrence of stroke within 90±7 days after administration | within 90±7 days
Changes in serum biomarkers (TNF-α, MMP9, CHE, IL-10, S100-β) from baseline on day 7 after administration | day 7

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: No